CLINICAL TRIAL: NCT01616446
Title: PHARMACOKINETICS OF CYCLOSPORIN - A MICROEMULSION IN CHILDREN WITH IDIOPATHIC NEPHROTIC SYNDROME
Brief Title: Pharmacokinetics of Cyclosporin in Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciana dos Santos Henriques, principal investigator, University of Sao Paulo
Other Study IDs: CLINICS-D-12-00179R1
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Nephrotic Syndrome
Keywords: cyclosporin; nephrotic syndrome; pharmacokinetics; children
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- remission: Nephrotic patients in remission
- relapse: Nephrotic patients in recidive

SUMMARY:
The purpose of this study is to evaluate whether there are differences in the pharmacokinetics of cyclosporine in remission nephrotic syndrome compared to relapsed disease in children.

DETAILED DESCRIPTION:
This is a prospective study on ten children using Cyclosporin-A (CSA) microemulsion to treat idiopathic nephrotic syndrome (INS), with normal renal function, who achieved complete remission with CSA. The objective is to compare the pharmacokinetic (PK) parameters of CSA in INS during remission and relapse of the disease. The PK profile of CSA was evaluated with the 12-hour area under the time-concentration curve (AUC0-12) using seven time-point samples. This procedure was done on each patient during remission and relapse with the same CSA dose in mg/kg/day. The AUC0-12 was calculated by trapezoidal rule. All PK parameters and the resumed 4-hour area under the time-concentration curve (AUC0-4) were correlated with AUC0-12. This study is very important because the cyclosporin is a nephrotoxic drug with narrow therapeutic window.

ELIGIBILITY:
Inclusion Criteria:

* children with steroid-resistant nephrotic syndrome and steroid-dependent nephrotic syndrome in use of cyclosporine
* renal function evaluated by creatinine clearance estimated by stature ≥ 90 ml/min/1.73m2
* cyclosporine trough level (C0) between 50 and 150 ng/ml
* complete remission with cyclosporine according to the guidelines of International Society of Kidney Diseases in Children

Exclusion Criteria:

* renal and hepatic function abnormalities
* presence of infectious disease
* clinical or histological signs of CSA nephrotoxicity and suspicious of non-compliance

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Iidiopathic nephrotic syndrome followed in the Pediatric Nephrology Unit of Instituto da Criança-HCFMUSP
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Henriques Ldos S, Matos Fde M, Vaisbich MH. Pharmacokinetics of cyclosporin--a microemulsion in children with idiopathic nephrotic syndrome. Clinics (Sao Paulo). 2012 Oct;67(10):1197-202. doi: 10.6061/clinics/2012(10)12. PMID 23070347